CLINICAL TRIAL: NCT02815306
Title: Polyaxial Brace Fixing for the Treatment of Congenital Clubfoot in Newborns and Infants
Brief Title: Polyaxial Brace Fixing for the Treatment of Congenital Clubfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Guoxin Nan, Chief of the orthopeadic deapartment, Children's Hospital of Chongqing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Guoxin CFB-2016
Record Dates: First submitted 2016-03-24; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Clubfoot
Keywords: Congenital idiopathic clubfoot; Pirani score; infant; polyaxial brace
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brace goup (Experimental): The infants who were brace group treated by braces which were designed and made by us.
  Interventions: Device: Polyaxial brace

INTERVENTIONS:
Device: Polyaxial brace — The Polyaxial brace were made by a technician trained by the China National Disabled Persons Federation. For all patients, gypsum models were prepared first, and then braces were fabricated according to the models. The detailed technique was fully in accordance with the Ponseti method.

SUMMARY:
Congenital idiopathic clubfoot (CC) is the fifth most common congenital malformation in children. The Ponseti method is an effective protocol for treatment of congenital idiopathic clubfoot. Plaster is essential for the Ponseti treatment. This paper describes a new brace that can be used for the treatment of clubfoot in newborns and infants instead of plaster.

DETAILED DESCRIPTION:
Methods In the orthopedic department of our hospital, 38 infants and newborns, (57 feet) ,all the patients were under the age of 3 months with congenital clubfoot underwent polyaxial braces between Jan, 2011 to Oct ,2013. Polyaxial brace was used for the deformity correction. Then, during the following 1-3 years, the Dennis braces were used during the night in case of recurrence. Prospective follow-up for a mean duration of 25 months (range, 15-36months) was carried out. The efficacy of the treatment was assessed by Pirani's scoring system before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

0-6 months infants parents would like to cooperate with the doctors.

Exclusion Criteria:

over 6 months.

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
hindfoot | 1 month
  severity of the posterior crease, emptiness of the heel and rigidity of the equinus
midfoot | 1 month
  curvature of the lateral border of the foot, severity of the medial crease and position of the lateral part of the head of the talus

IPD SHARING:
Plan to Share IPD: Undecided